CLINICAL TRIAL: NCT02771301
Title: Safety and Efficacy of IDH1R132H-DC Vaccine in Gliomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Yanda Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Nan Ji, Professor of Neurosurgery, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDH1
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Glioma
Keywords: IDH1R132H Dendritic cell glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dendritic cell (Other): Patients will receive autolgous IDH1R132H dendritic cells and cytotoxic lymphocytes treatment.
  Interventions: Biological: dendritic cells

INTERVENTIONS:
Biological: dendritic cells — Concurrent of radiotherapy and chemotherapy plus 12 cycles of dendritic cells and cytotoxic lymphocytes treatment

SUMMARY:
This trial is aimed at evaluating the safety and efficacy of IDH1R132H-DC vaccine in glioma with IDH1R132H mutation.

DETAILED DESCRIPTION:
Eligible patients that provide written informed consent will undergo apheresis to collect blood mononuclear cells for vaccine production. All patients will receive mature dendritic cells for a total of 12 vaccine doses.The DC vaccine will be given subcutaneously every four weeks. Peripheral blood will be taken two weeks after injection each time to monitor the immune response.

ELIGIBILITY:
Inclusion Criteria:

* The patient signed "informed consent" voluntarily;
* The age of patient is between 18 and 70 years;
* The tumor can be resected and tumor resection rate ≥80%;
* IDH1R132H mutation can be confirmed by immunohistochemistry or real-time quantitative PCR;
* Peripheral blood lymphocytes absolute value is not less than 0.8 × 106;
* KPS score ≥70 ;
* The patient has normal bone marrow reserve and normal liver and kidney function ( The bone marrow, liver and kidney function must be confirmed by Laboratory examination to meet the requirements of participating in the study within 3 days before the first acceptance of IDH1R132H-DC tumor vaccine therapy): Medium neutrophil absolute value ≥1,500 / mm3; hemoglobin> 10g / dL; platelet count> 100,000 / mm3; total bilirubin <1.5 × ULN; alanine aminotransferase / aspartate aminotransferase <2.5 × ULN; serum creatinine <1.5 × ULN;
* Normal heart function ;
* Better follow-up and compliance;
* For women of childbearing age (15 to 49 years)，pregnancy test must be negative 7 days before starting this study. Male and female patients of childbearing potential must agree to use effective contraceptive measures to ensure that during the study period and three months after cessation of treatment will not be pregnant.

Exclusion Criteria:

* The patient did not sign "informed consent" or signed unvoluntarily.
* Non-glioma patients
* Drugs for brain or antibody therapy had been used 4 weeks before the start of this study
* Active infection
* Human immunodeficiency virus (HIV) positive
* Hepatitis C or hepatitis B infective
* Pregnancy or breast-feeding women
* Patients did not agree to use effective contraception during treatment and the following 3 months.
* Patients also participated in other clinical studies.
* The subjects researchers believe are not suitable for participation or completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Efficacy of IDH1R132H dendritic cell vaccine as measured by adverse events | 2 year
  2 years progress free survival and overall suvival as measured by RECIST criteria 4.0

SECONDARY OUTCOMES:
Antigen specific cell responses before and after vaccination | 2 year
  Immunological response based on measuring increased numbers of IDH1R132H specific T cells and levels of anti-IDH1R132H antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Ji, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Hebei Yanda Hospital, Sanhe, Hebei

IPD SHARING:
Plan to Share IPD: Undecided